CLINICAL TRIAL: NCT02665637
Title: A Randomized, Double-blind, Two-arm, Parallel-group, Single Dose Study to Compare the Pharmacokinetics, Safety and Immunogenicity of Two Formulations of Trastuzumab (CT-P6 and US-licensed Herceptin) in Healthy Subjects
Brief Title: Study Comparing Pharmacokinetics, Safety and Immunogenicity of CT-P6 and US-licensed Herceptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CT-P6 1.5
Record Dates: First submitted 2016-01-12; First posted 2016-01-28 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P6 (Active Comparator): Trastuzumab
  Interventions: Drug: Trastuzumab
- US-licensed Herceptin (Active Comparator): Trastuzumab
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Each patient may receive single dose by intravenous infusion

SUMMARY:
This is a double-blind, two-arm, parallel-group, single-dose study.

DETAILED DESCRIPTION:
This is a double-blind, two-arm, parallel-group, single-dose study. A total of 70 healthy male subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject
2. Subject voluntarily agrees to participate in this study

Exclusion Criteria:

1. Female.
2. Subject has a medical condition of disease including one or more.
3. Smoker

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics will be assessed by AUC | up to week 10
  Pharmacokinetics will be assessed by AUC.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wood-Horrall, MD, Principal Investigator — PPD Phase I Clinic
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States